CLINICAL TRIAL: NCT06049264
Title: Short-term Effects of Thoracic Spine Manual Traction With Mobilization Versus Thoracic Manipulation in Patients With Mid Thoracic Pain and Pseudo Visceral Symptoms
Brief Title: Thoracic Spine Manual Traction With Mobilization Versus Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0132 Feroza
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Thoracic
Keywords: Manipulation; Mobilization; Pseudo visceral symptoms; Pain; Spinal Traction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Spine Manual Traction with Mobilization (Experimental): Thoracic Spine Manual Traction with Mobilization
  Interventions: Other: Thoracic spine manual traction with mobilization protocol.
- Thoracic Spine Manual Traction with Manipulation (Active Comparator): Thoracic Spine Manual Traction with Manipulation
  Interventions: Other: Thoracic manipulation protocol

INTERVENTIONS:
Other: Thoracic spine manual traction with mobilization protocol. — The therapist will perform one 30-second bout of grade I or II central posterior-anterior mobilization at the T3 spinous process as described by Maitland et al. After the 30-second bout, the therapist proceeded to T4 and performed the same technique. This process was continued sequentially in a caudal direction to T8, for an overall intervention time of approximately 3 minutes. In addition to mobilization, thoracic spine traction will be also given in sitting position.
  Arms: Thoracic Spine Manual Traction with Mobilization
Other: Thoracic manipulation protocol — To perform the manipulation, the stabilizing hand will be placed at the level immediately caudal to the restricted segment using a ''pistol grip''. Once the pre manipulative position will be achieved the patient will be instructed to take a deep inhalation and exhale. During the exhalation the treating clinician performed a high velocity, small amplitude thrust in a direction to facilitate relative closing or opening of the respective facet joint as indicated by the segmental examination.
  Arms: Thoracic Spine Manual Traction with Manipulation

SUMMARY:
This project will be a Randomized clinical trial conducted to compare Short-term effects of thoracic spine manual traction with mobilization and Thoracic manipulation in patients with mid thoracic pain and pseudo visceral symptoms. Sample will be collected through non-probability convenient sampling, following eligibility criteria from Sehat Medical complex, Lahore. Eligibility criteria will be Age group between 20 to 40 years both male and female genders with mid thoracic pain having pseudo visceral symptoms. Referred by physician after exclusion of post-surgical condition from past 6 months Neurological, Pulmonological, Cardiac, Musculoskeletal and Esophageal conditions. Participants will be randomly allocated in two groups via sealed envelope method, baseline assessment will be done, Group A participants will be given baseline treatment along with Thoracic spine manual traction with mobilization, Group B participants will be given baseline treatment along with Thoracic manipulation protocol. Pre and post intervention assessment will be done via, Numeric pain rating scale(NPRS), Revised Oswestry thoracic pain disability questionnaire (ODI) and Inclinometer to measure ROM of Thoracic spine,3 sessions per week will be given for 4 weeks, data will be analyzed by using SPSS version 29.

DETAILED DESCRIPTION:
Spinal pain is a well-recognized condition associated with significant personal and community burdens. Compared to the lumbar and cervical spine, the thoracic spine has received less attention in terms of clinical, genetic and epidemiologic research, yet pain experienced in the thoracic spine can be equally disabling, imposing similar burdens on the individual, community and workforce. Pseudo visceral symptoms refer to physical sensations or symptoms that mimic those associated with underlying medical condition affecting the internal organs, but without any organic cause or pathology. Manipulation and mobilization are two manual techniques that are commonly used by osteopaths, chiropractors and physiotherapists to treat spinal pain and dysfunction. This study aims to compare Short-term effects of thoracic spine manual traction with mobilization and Thoracic manipulation in patients with mid thoracic pain and pseudo visceral symptoms.

This randomized clinical trial will be conducted at Sehat medical complex, Lahore. It will include patients with age group between 20 to 40 years, both male and female gender with mid thoracic pain and pseudo visceral symptoms referred by physician after exclusion of visceral symptoms. Those patients with post-surgical condition from past 6 months, Neurological, Pulmonological or Cardiac conditions will be excluded. Participants will be divided into two groups. Group A will receive of thoracic spine manual traction with mobilization treatment protocol and Group B will receive Thoracic manipulation protocol. Both groups will receive baseline treatment including TENS and Hot pack. Short term effects would be assessed after treatment for 4 weeks. Patients will be assessed by Numeric pain rating scale, Inclinometer and Revised Oswestry thoracic pain disability questionnaire. The findings can contribute to the growing evidence based supporting whether the use of thoracic spine manual traction with mobilization or Thoracic manipulation improve pain, ROM and disability in patients with mid thoracic pain and pseudo visceral symptoms. Analysis will be done by statistical package for social sciences SPSS 29.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 20 to 40 years
* Both male and female gender.
* Mid thoracic pain with pseudo visceral symptoms.
* Participants with moderate and severe pain as ODI score should be within range of 30% to 68%.
* Referred by physician after exclusion of visceral symptoms

Exclusion Criteria:

* Post-surgical condition (6 months)
* Neurological Conditions
* Pulmonological conditions
* Cardiac conditions such as angina pectoris, coronary artery disease, Arrhythmia, pericarditis or aortic aneurysm.
* Musculoskeletal disorders
* Esophageal disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4th Week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
Revised Oswestry thoracic pain disability questionnaire for disability | 4th Week
  This questionnaire is designed to evaluate Level of Disability in thoracic Pain patients. Disability was measured using the Oswestry Disability Index (ODI: range 0-no disability to 50-maximum disability possible). The ODI is a commonly used outcome measure amongst LBP patient.
Inclinometer measurement of Thoracic ROM | 4th Week
  Inclinometers are portable, lightweight, and inexpensive pieces of equipment that are used to measure range of motion, like goniometry. Inclinometers are typically found in clinics and are used as a part of a physical examination. An intraclass correlation coefficient (ICC) was found to be between 0.87-0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Sehat Medical Complex, Hanjarwal Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izzo R, Popolizio T, D'Aprile P, Muto M. Spinal pain. Eur J Radiol. 2015 May;84(5):746-56. doi: 10.1016/j.ejrad.2015.01.018. Epub 2015 Feb 13. PMID 25824642
- [Background] Briggs AM, Smith AJ, Straker LM, Bragge P. Thoracic spine pain in the general population: prevalence, incidence and associated factors in children, adolescents and adults. A systematic review. BMC Musculoskelet Disord. 2009 Jun 29;10:77. doi: 10.1186/1471-2474-10-77. PMID 19563667
- [Background] Romanchuk O. The Immediate Effects of the Manual Therapy Traction Manipulations on Parameters of Cardiorespiratory System Functioning. International Journal of Human Movement and Sports Sciences. 2022;10(4):832-40.
- [Background] Morningstar MW. Cervical hyperlordosis, forward head posture, and lumbar kyphosis correction: A novel treatment for mid-thoracic pain. J Chiropr Med. 2003 Summer;2(3):111-5. doi: 10.1016/S0899-3467(07)60055-X. PMID 19674605
- [Background] Manchikanti L, Singh V, Pampati V, Beyer CD, Damron KS. Evaluation of the prevalence of facet joint pain in chronic thoracic pain. Pain Physician. 2002 Oct;5(4):354-9. PMID 16886012
- [Background] Takatalo J, Ylinen J, Pienimaki T, Hakkinen A. Intra- and inter-rater reliability of thoracic spine mobility and posture assessments in subjects with thoracic spine pain. BMC Musculoskelet Disord. 2020 Aug 10;21(1):529. doi: 10.1186/s12891-020-03551-4. PMID 32778081
- [Background] Cleland JA, Flynn TW, Childs JD, Eberhart S. The audible pop from thoracic spine thrust manipulation and its relation to short-term outcomes in patients with neck pain. J Man Manip Ther. 2007;15(3):143-54. doi: 10.1179/106698107790819828. PMID 19066662
- [Background] . Fryer G, Carub J, McIver S. The effect of manipulation and mobilisation on pressure pain thresholds in the thoracic spine. Journal of Osteopathic Medicine. 2004;7(1):8-14.
- [Background] Vicenzino B, Collins D, Wright A. The initial effects of a cervical spine manipulative physiotherapy treatment on the pain and dysfunction of lateral epicondylalgia. Pain. 1996 Nov;68(1):69-74. doi: 10.1016/S0304-3959(96)03221-6. PMID 9252000
- [Background] Park SJ, Kim SH, Kim SH. Effects of Thoracic Mobilization and Extension Exercise on Thoracic Alignment and Shoulder Function in Patients with Subacromial Impingement Syndrome: A Randomized Controlled Pilot Study. Healthcare (Basel). 2020 Sep 2;8(3):316. doi: 10.3390/healthcare8030316. PMID 32887287
- [Background] Anandkumar S M Sc Pt Bpt C-Ompt Cafs Cert Dnt, Manivasagam M Bpt Dyt Comt Fsr Dnp Ces. Effect of fascia dry needling on non-specific thoracic pain - A proposed dry needling grading system. Physiother Theory Pract. 2017 May;33(5):420-428. doi: 10.1080/09593985.2017.1318423. Epub 2017 May 8. PMID 28481688